Effect of Unilateral Ultrasound-Guided Subcostal Transversus Abdominis Plane Block in Patients Undergoing Laparoscopic Sleeve Gastrectomy

PI: Christina Jeng, MD NCT03856788

Document Date: Aug 24, 2022

Statistical Analysis Plan

Baseline descriptive statistics will be performed for demographic variables, intraoperative data, and for potential confounders. All variables will be checked for normality via Kolmogorov–Smirnov test or Shapiro–Wilk test as well as histogram visual inspection. Normal variables will be reported as mean, standard deviation, non normal variables will be reported as median [IQR]. Proportions will be reported as n(%) and analyzed via Chi Square test. Normal continuous variables will be analyzed via t test, or paired t-test depending on the variable. Non-non normal variables will be tested via Mann-Whitney U test. Area-under the curve analyses will be evaluated through ROC analysis or other tests as indicated. Where applicable, linear or logistic regression will be utilized to assess for associations of variables for both univariate and multivariate analysis.